CLINICAL TRIAL: NCT06978530
Title: Mandibular Sub-condylar Fractures Fixation Using Three-dimensional Custom Plate Versus Standard Titanium Fixation Plates: Randomized Clinical Trial
Brief Title: 3D Custom Plate vs. Standard Titanium Plates for Mandibular Sub-condylar Fractures Fixation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esraa Mosad Tawfik (Other)
Responsible Party: Sponsor-Investigator, Esraa Mosad Tawfik, Resident, Oral and Maxillofacial Surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D-SCF-RCT-2025
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mandibular Sub-condylar Fracture
Keywords: Mandibular fracture; 3D custom plate; titanium miniplates; sub-condylar fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Custom Plate group (Experimental): Patients in this group will undergo open reduction and internal fixation of displaced mandibular sub-condylar fractures using preoperatively designed and 3D-printed patient-specific titanium plates.
  Interventions: Device: 3D custom plate
- Standard titanium plates group (Active Comparator): Patients in this group will undergo open reduction and internal fixation of displaced mandibular sub-condylar fractures using the conventional technique, involving either two standard titanium miniplates or a single 2.3 mm titanium plate.
  Interventions: Device: Standard titanium fixation plates

INTERVENTIONS:
Device: 3D custom plate — Custom 3D plate will be designed using preoperative CT and virtual surgical planning.
  Other Names: patient specific plate
  Arms: 3D Custom Plate group
Device: Standard titanium fixation plates — The fixation will be performed according to established surgical principles for managing displaced mandibular sub-condylar fractures without patient-specific planning or customization.
  Arms: Standard titanium plates group

SUMMARY:
This randomized clinical trial aims to conduct a comprehensive clinical and radiographic evaluation by comparing the efficacy of standard titanium fixation plates with three dimensional custom plate in the management of sub-condylar fractures. By assessing the clinical outcomes, accuracy of reduction of the fracture segments, and bite force promoted by both fixation modalities.

ELIGIBILITY:
Inclusion Criteria:

* Displaced sub condylar fractures, requiring open reduction and rigid internal fixation
* Age ranges from 18 to 60 years
* Fracture duration less than 2 weeks
* Patients with adequate follow up duration for outcome assessment

Exclusion Criteria:

* Comminuted sub condylar fractures
* Patients with severe systemic diseases that may affect fracture healing
* Presence of any pathology at the fracture site
* Patients with previous history of mandibular surgery
* Medically compromised patients who are not fit to undergo surgery under general anesthesia
* Patients with in complete medical records or missing follow up data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Bite force | 1 month, 3 months, and 6 months postoperatively
  Bite force measured in Newtons at the molar region using a bite force recording device.

SECONDARY OUTCOMES:
Maximum mouth opening | 1 month, 3 months, and 6 months postoperatively.
  Distance in mm between incisal edges during maximal mouth opening.
Mandibular deviation on opening | 1 month, 3 months, and 6 months postoperatively.
  Deviation in mm measured using midline reference.
Accuracy of fracture reduction | Immediately postoperative (within 1 week)
  Evaluated by comparing preoperative CT with postoperative CT using 3D image superimposition analysis